CLINICAL TRIAL: NCT06134856
Title: Quantitative Sensory Testing Changes Following Talocrural Joint Manipulation in People With Achilles Tendinopathy; A Randomized Controlled Trial
Brief Title: A Study Examining Changes in Pain After Manual Therapy in People With Achilles Tendon Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philadelphia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC02117
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-08

CONDITIONS: Achilles Tendinopathy; Ankle Strain; Achilles Tendon Pain; Achilles Tendonitis
Keywords: Achilles; Tendinopathy; Tendonitis; Ankle; Pain
MeSH Terms: conditions — Tendinopathy; Pain

STUDY DESIGN:
Intervention Model Description: Randomized control trial, treatment group and control group
Who Masked: Participant
Masking Description: Subjects in the control group will receive 1 minute of passive ankle movement into ankle dorsiflexion. The researcher will not move the subject's ankle into a point where tissue stretch/tension is perceived. This will serve as an appropriate sham treatment since it still involves the subjects perception of treatment and includes the hands-on element of manual therapy, without the use of any tissue intervention which would theoretically effect change.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Subjects assigned to the intervention group will then receive a talocrural joint high velocity, low amplitude thrush mobilization/manipulation. Standardized technique for this procedure involves the subject long-sitting with their back supported on the treatment table. The provider will then passively dorsiflex and evert the ankle to the point at which a joint tension end-feel is obtained.
  A small amplitude of movement is rapidly provided by the provider in a caudal direction. The provider may attempt up to three treatment thrust impulses, or until an audible cavitation is heard, indicating joint movement. Even without an audible cavitation, no more than three impulses will be provided. Some research in other body regions indicates that treatment effect is present even in those with whom audible joint cavitation is not noted.
  Interventions: Procedure: Ankle mobilization
- Control (Sham Comparator): Subjects in the control group will receive 1 minute of passive ankle movement into ankle dorsiflexion. The researcher will not move the subjects ankle into a point where tissue stretch/tension is perceived. This will serve as an appropriate sham treatment since it still involves the subjects perception of treatment and includes the hands-on element of manual therapy, without the use of any tissue intervention which would theoretically effect change.
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Procedure: Ankle mobilization — Ankle joint mobilization as described in treatment arm description
  Arms: Intervention
Procedure: Sham treatment — Light passive movement of the foot and ankle, avoiding the end-ranges which may actually elicit a mechanical change
  Arms: Control

SUMMARY:
The purpose of this research is to find out how pain sensation may change in the Achilles tendon after the use of manual physical therapy. The testing itself will use a device that gradually produces a sensation of heat or cold on your skin, which we will place directly over your Achilles Tendon. You will let the researcher know when the heat or cold becomes what you would describe as "slight discomfort," at which point the pressure will be stopped. Testing will be completed three (3) times in a row. The device has built-in programming which ensures that the heat or cold applied will be safe, even though it may be briefly uncomfortable. After this first testing the researchers will perform 1-3 repetitions of the ankle joint mobilization/manipulation. This technique involves the researcher providing a small quick stretching movement downwards at the ankle. This is a common therapeutic technique utilized by Physical Therapists, chiropractors, and physicians and is considered very safe. After this treatment we will perform the same measurements of hot and cold discomfort on your Achilles tendon

DETAILED DESCRIPTION:
While healthcare's understanding of sensory processing changes has grown significantly in the last several years, numerous gaps in the literature exist. In particular, lower extremity tendinopathies, while common, have not been well studied through the lens of potential sensory sensitizations. The prevalence of Achilles Tendinopathy has been reported to be around 6%, meaning that Millions of individuals in the United States will have these issues at any given time. Historically, clinical management of the condition has been challenging. This study aims to provide data for clinicians to better inform treatment strategies by increasing knowledge of the neurosensory changes that may accompany the condition.

After subjects complete informed consent, they will then answer a brief intake screening form asking for demographic information and symptom history to confirm eligibility. The clinical screening will then be performed to confirm signs of Achilles tendinopathy, namely assessment for tenderness to palpation in the Achilles Tendon, the the Royal London Hospital Test. The Royal London Hospital Test consists of assessing for tenderness in the Achilles tendon with the ankle in a relaxed position, and then again with the subject in maximal active dorsiflexion. A positive test is noted when tenderness is reduced in the maximally dorsiflexed position as compared to the rest state. Once eligibility is confirmed, a subject number will be assigned. Prior to beginning data collection, a random number generation program will be used to determine which subject numbers will be placed into the intervention and control groups. All participants will begin data collection with standardized assessment of heat and cold pain thresholds. Heat and cold pain threshold testing will be performed using the Medoc TSA Air2, with calibration performed before each data collection session. Data collection will be performed in accordance with the protocols set forth by the German Research Network on Neuropathic Pain (DFNS.) Participants will be instructed to press the input button to stop the trial when the heat or cold pain stimulus becomes what each subject would describe as pain or discomfort.

Subjects will be instructed that it is a threshold test, not a tolerance test, thus they are asked to press the stop trial button at the beginning of pain, not at their maximal tolerable amount. All trials will be completed three times with a pre-determined 15 second rest between trials. All three trials will be averaged for data analysis purposes. Subjects assigned to the intervention group will then receive a talocrural joint high velocity, low amplitude thrush mobilization/manipulation. Standardized technique for this procedure involves the subject long-sitting with their back supported on the treatment table. The provider will then passively dorsiflex and evert the ankle to the point at which a joint tension end-feel is obtained.

A small amplitude of movement is rapidly provided by the provider in a caudal direction. The provider may attempt up to three treatment thrust impulses, or until an audible cavitation is heard, indicating joint movement. Even without an audible cavitation, no more than three impulses will be provided. Some research in other body regions indicates that treatment effect is present even in those with whom audible joint cavitation is not noted. (10) Subjects in the control group will receive 1 minute of passive ankle movement into ankle dorsiflexion. The researcher will not move the subject's ankle into a point where tissue stretch/tension is perceived. This will serve as an appropriate sham treatment since it still involves the subjects perception of treatment and includes the hands-on element of manual therapy, without the use of any tissue intervention which would theoretically effect change.

Immediately following the application of the intervention or sham all participants will be re-tested for heat and cold pain thresholds in the same manner utilized at baseline. For ethical purposes, subjects assigned to the control group will also receive the intervention following data collection.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who self-report pain in the back of the heel (Achilles tendon) persisting for at least 3 months.

Prior to inclusion in the study, subjects will undergo a brief clinical screen by the investigators to confirm the signs of Achilles tendinopathy. This screen will consist of assessing for tenderness to palpation in the Achilles tendon and the Royal London Hospital Test (Tenderness to pressure is assessed with the subject in maximal active dorsiflexion and is positive if reduced in this position as compared to the resting state.)

Exclusion Criteria:

* History of any surgery distal to the fibular head on the involved lower extremity
* Cortisone injection to the painful Achilles tendon within the last 6 months
* History of diagnosed ankle joint or connective tissue instability
* Current pregnancy
* Age under 18 years of age
* Unable or unwilling to give consent for test and/or treatment procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Heat and Cold Thresholds | Baseline and 1 hour
  Outcome variables will be mean scores for 3 trials each of heat and cold pain threshold, measured in degrees centigrade, initially and immediately (within 5 minutes) after the intervention or sham intervention, with analysis of threshold change measured in the post-test as compared to the baseline data.

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Lowe, Principal Investigator — PCOM
Locations (1):
- Philadelphia College of Osteopathic Medicine-GA, Suwanee, Georgia, United States

IPD SHARING:
Plan to Share IPD: No